CLINICAL TRIAL: NCT05500612
Title: Magnetic Resonance Imaging of Hypoxia for Radiation Treatment Guidance in Glioblastoma Multiforme (MANGO)
Brief Title: MRI Hypoxia Study for Glioblastoma Multiforme (GBM) Radiation Therapy
Acronym: MANGO
Status: Not yet recruiting | Type: Observational
Sponsor: University of Sydney (Other)
Collaborators: The Brain Cancer Group (Unknown)
Responsible Party: Sponsor
Other Study IDs: ETH11794
Record Dates: First submitted 2022-08-09; First posted 2022-08-15 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is designed to evaluate the role of Oxygen Enhanced (OE) Magnetic resonance imaging (MRI) and Blood Oxygenation Level Dependent (BOLD) MRI in detecting regions of hypoxic tumour and to evaluate their use as imaging methods to selectively deliver targeted radiotherapy to regions of aggressive disease.

DETAILED DESCRIPTION:
The ability to image tumour hypoxia at diagnosis and prior to radiotherapy is extremely important to appropriately adapt radiotherapy plans such that to selectively deliver higher doses of radiation to those more aggressive tumour subregions, thereby improving the chances to achieve better local tumour control. Preoperative imaging of tumour hypoxia also offers the opportunity for 'supra-marginal resections' in surgical planning beyond current neurosurgical standard of care. Additionally, accurately identifying regions of tumour hypoxia harbouring tumour progression at follow up is fundamental in patient follow-up, allowing multidisciplinary teams to more confidently intervene at an earlier stage of tumour recurrence and personalise therapy tailored to the tumour's response to treatment. Routine imaging of tumour hypoxia is currently challenging, as it requires [18F]-Fluoromisonidazole (18F-FMISO PET) imaging, which is not available in the majority of clinical centres. Today, the availability of accelerated quantitative MRI sequences on clinical MRI systems could enable quantification of tumour hypoxia without putting an unfeasible burden on patients' scan sessions. The next frontier in radiotherapy treatment will use these techniques to identify hypoxic tumour tissues and personalise treatments to the patient's unique tumour biology, maximising the probability of tumour control.

This clinical study will acquire additional images of brain cancer patients. The images will not change the patient's treatment. This study is designed to evaluate the role of oxygen enhanced (OE) MRI and BOLD MRI in detecting regions of hypoxic tumour and to evaluate their use as imaging methods to selectively deliver targeted radiotherapy to regions of aggressive disease.

ELIGIBILITY:
Inclusion Criteria:

* Suspected high-grade glioma (HGG) / glioblastoma multiforme (WHO grade IV) at initial radiological examination
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2
* Available for scanning on two separate days

Exclusion Criteria:

* Women lactating, pregnant or of childbearing potential who are not willing to avoid pregnancy during the study
* Patients with a history of severe renal disease(s) (eGFR <20) that cannot tolerate gadolinium chelate contrast agents.
* Geographically remote patients unable to agree to imaging schedule
* Patients who have received anti - vascular endothelial growth factor (anti-VEGF) monoclonal antibody therapy the 3 months prior to recruitment
* Patients with a history of psychological illness or condition such as to interfere with the patient's ability to understand the requirements of the study.
* Patients with significant cardiac or pulmonary disease including cardiac arrythmias or Chronic Obstructive Pulmonary Disease (COPD) that are unable to tolerate high flow O2 for oxygen contrast.
* Patients taking carbonic anhydrase inhibitors (Acetazolamide)
* History of glaucoma
* Any implant, foreign body, 3 Tesla (3T) MRI incompatible device, or other contraindication to MRI imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histopathological diagnosis of a high grade glioma / glioblastoma multiforme
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Determination of spatial correlation of hypoxic tumour volume between Magnetic resonance imaging (MRI) and [18F]-Fluoromisonidazole (18F-FMISO) MRI | 1 year
  Spatial correlation between hypoxic tumour volume determined with MRI and 18F-FMISO will be evaluated via measurements of Dice similarity coefficient. Dice similarity coefficients > 0.9 will be considered a strong spatial correlation. Quantitative correlation of voxel-wise levels of hypoxia will be evaluated via measurement of the Spearman's/Pearson's correlation coefficient. Correlation coefficients > 0.7 will be considered a strong correlation.

SECONDARY OUTCOMES:
Repeatability of voxel-wise levels of hypoxia in the tumour | 1 year
  Repeatability of voxel-wise levels of hypoxia in the tumour will be assessed by measurements of intraclass correlation coefficient (ICC).27 ICC values > 0.9 reflect excellent repeatability, good between 0.75 and 0.9, moderate between 0.5 and 0.75, and poor < 0.5. Additionally, similarity between the hypoxia tumour volume (HTV) defined with the MRI biomarker at the two timepoints will be assessed via calculation of Dice similarity coefficient. Dice similarity coefficients > 0.9 will be considered a strong correlation.
The predicted patient outcomes of the biologically-adapted Radiotherapy (RT) plan will be compared with the actual patient outcomes | 1 year
  The predicted patient outcomes of the biologically-adapted RT plan will be compared with the actual patient outcomes following conventional treatment, by using metrics including tumour control probability (TCP) and toxicity measurement to organs at risks and healthy brain (including equivalent uniform dose). Success for this objective will be achieved if the biologically-adapted RT plans result in improved TCP by at least 10% for all patients over conventional treatment, while toxicity metrics remain similar.
Correlation between the percentage of hypoxic tumour volume and clinical outcome | 1 year
  Correlation between the percentage of hypoxic tumour volume and clinical outcome will be evaluated by means of hazard ratio obtained from Cox regression. A hazard ratio > 1 (p<0.05) will indicate that the hypoxic tumour volume increase from 13 weeks post chemoradiation therapy (CRT) and recurrence is associated with worst Overall Survival (OS) and Progression Free Survival (PFS).
Correlation between the percentage change of hypoxic tumour volume during treatment and clinical outcome | 1 year
  Correlation between the percentage change of hypoxic tumour volume during treatment and clinical outcome will be evaluated by means of hazard ration obtained from Cox regression. A hazard ratio > 1 (p<0.05) will indicate that the increase in hypoxic tumour volume during treatment is associated with worse OS.

CONTACTS AND LOCATIONS:
Overall Officials: Caterina Brighi, Principal Investigator — University of Sydney
Locations (2):
- Australia (2):
  - North Shore Private Hospital, St Leonards, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales

IPD SHARING:
Plan to Share IPD: Yes
After study completion, de-identified (non-coded, non-re-identifiable) data will be available to researchers for further scientific research. Information about data sharing will be provided to study participants in the Patient Information Sheet.
Supporting Information: Study Protocol, ICF
Time Frame: After study completion.
Access Criteria: Data stored at the university: In order to download / decompress the stored, de-identified data, participating researchers will agree to the terms of use for the data, including that the data are not to be published or otherwise redistributed without the express consent of the original investigator(s).
  Data stored at an external repository: de-identified study data may be provided to an external research data repository, archive or register so that it may be made publicly available for other scientific research. Study data that are provided to an external research data repository will be stored at and managed by the external repository. Data will only be shared with repositories whose function has been reviewed and approved by an accredited Research Integrity/Ethics Committee/Board, under a Materials Transfer Agreement with the University.